CLINICAL TRIAL: NCT05592977
Title: Effect of Bilateral Distalization of Upper First Molars in a Group of Patients After Extraction of Maxillary Second Molars Using Infra Zygomatic Mini Implants: A Prospective Clinical Trial
Brief Title: Effect of Bilateral Distalization of Upper First Molars in a Group of Patients After Extraction of Maxillary Second Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Hosam Abdullah Mohamed Zaza, Principle investigator, Future University in Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUE.REC(23)/11-2020
Record Dates: First submitted 2021-06-05; First posted 2022-10-25 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Class II Malocclusion
Keywords: Intermolar Width; Molar Inclination; Intra-oral Appliance; Infrazygomatic Mini-screws; Distalization
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Masking Description: Due to the nature of the study, the operator and patients can't be blinded. Blinding of the outcome assessors can be done by sealing the name of the patient in the pre and post treatment radiographs used for analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-oral Distalizing Appliance (Experimental): Two infra zygomatic mini-implants will be placed Bands will be cemented to upper first molars. The inner bow (1.2mm) is a modified version of the inner part of a conventional face bow. Two hooks were soldered onto the inner bow distal to the lateral incisor teeth regions, and U loop at 1st premolar region, and bends acting as mesial stop will be bent in front of the maxillary first molars.
  Orthodontic force 300 mg per side Will be delivered by Niti closed coil spring which is attached from infra zygomatic mini screw to the hook soldered to the wire framework.
  Interventions: Device: Intra-Oral Distalizing Device

INTERVENTIONS:
Device: Intra-Oral Distalizing Device — The inner bow (1.2mm) is a modified version of the inner part of a conventional face bow. Two hooks were soldered onto the inner bow distal to the lateral incisor teeth regions, and U loop at 1st premolar region, and bends acting as mesial stop will be bent in front of the maxillary first molars. The anterior component of the inner bow is 3 mm free from the labial surface of anterior teeth

SUMMARY:
There is a scarcity in the current literature regarding such appliance and its effect on distalizing the first maxillary molar in absence of the second molar. Therefore, this study was made to evaluate the effect of bilateral distalization of upper first molars in a group of patients after extraction of maxillary second Molars using infra zygomatic mini implants.

DETAILED DESCRIPTION:
The appliances available for distalization used to be mainly extraoral distalizing appliances which depended entirely on patient cooperation and compliance. Even after the emergence of intra-oral distalizing appliances they had adverse dentoalveolar effect such as anchorage loss and flaring of the upper anterior teeth. Thus, this study was made in order to evaluate the efficiency of our proposed appliance in the treatment of Class II patients while avoiding the adverse effects mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients with cervical vertebra maturation index (CVMI) 5 & 6.
* From quarter unit to 3\4-unit class II molar relationship.
* An overjet of an average 6mm.
* Full Set of permanent dentition except for the maxillary second molar.
* Favorable path of eruption for the maxillary third molar.

Exclusion Criteria:

* Medically compromised Patients.
* Patients under long term medications.
* Patients having sever periodontal disease.
* CVMI 3 or less
* Full unit class II cases

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
linear distalization of maxillary 1st molar. | Up until Class I Molar Relation (a maximum of 8 months regardless)
  Efficiency of the proposed appliance to induce distalization of the upper 1st molar measured on Scanned dental casts as well as cone-beam computed tomography (CBCT) in millimetres.
Rate of maxillary 1st molar Distalization in mm/ month. | Up until Class I Molar Relation (a maximum of 8 months regardless)
  Efficiency of the proposed appliance to induce distalization of the upper 1st molar measured on Scanned dental casts with a monthly follow up in millimetres.

SECONDARY OUTCOMES:
Changes in Intermolar width in mm. | Up until Class I Molar Relation (a maximum of 8 months regardless)
  Effect of the proposed appliance on the transverse Dental changes in the upper buccal segment through scanned dental cast in millimetres
Changes of Molar inclination in degrees. | Up until Class I Molar Relation (a maximum of 8 months regardless)
  Effect of the proposed appliance on the angulation of the first permanent molar through scanned dental cast and cone-beam computed tomography (CBCT) in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Mostafa, Professr and Chairman, Study Director — Future University in Egypt
Locations (1):
- Future University In Egypt, New Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD)
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available after publication

DOCUMENTS (2):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT05592977/Prot_000.pdf
  • Informed Consent Form (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT05592977/ICF_001.pdf